CLINICAL TRIAL: NCT06612047
Title: Comparison of 5.0T and 3.0T Biparametric Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer: A Prospective, Single Center and Paired-design Diagnostic Study
Brief Title: Comparison of 5.0T and 3.0T Biparametric Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer
Acronym: 5TbpMRI
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, XiaoJun, Professor, Chief Physician, Anhui Provincial Hospital
Other Study IDs: 2024-ky399
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; prostate biospy; Biparametric Magnetic Resonance; Prostate Imaging-Reporting and Data System; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinical suspicion of prostate cancer undergo 5.0T and 3.0T bpMRI: All enrolled patients need to undergo 5.0TbpMRI and 3.0TbpMRI (within one month). The magnetic resonance imaging sequences mainly include T1WI, multi-plane T2WI and multi-b-value DWI images.
  Interventions: Procedure: Prostate biopsy

INTERVENTIONS:
Procedure: Prostate biopsy — All patients were required to underwent transperineal prostate biopsy (Systemetic + Targeted) and have corresponding pathological diagnosis results.

SUMMARY:
The goal of this observational study is to compare 5.0T and 3.0T biparametric magnetic resonance imaging in the diagnosis of prostate cancer. The main aims of this study are:

* Compare the diagnostic efficacy of 5.0TbpMRI and 3.0TbpMRI for prostate cancer. Preliminarily evaluate the value of 5.0TbpMRI in diagnosing prostate cancer.
* Compare and analyze the accuracy of 5.0TbpMRI and 3.0TbpMRI in determining the T stage of prostate cancer. Preliminary evaluation of the value of 5.0TbpMRI in determining the tumor stage of prostate cancer.

The data of participants was collected prospectively.

DETAILED DESCRIPTION:
The methods currently recommended by the guidelines for early diagnosis of prostate cancer mainly include rectal examination, serum prostate-specific antigen detection, transrectal prostate ultrasound, and multi-parameter magnetic resonance imaging. However, these methods lack sufficient specificity for the diagnosis of prostate cancer. Therefore, prostate biopsy is still the gold standard for the diagnosis of prostate cancer. mpMRI has good accuracy in detecting clinically significant prostate cancer, but mpMRI is difficult to identify lesions with a tumor diameter of less than 5 mm, and false positive results may occur for benign diseases such as prostatitis. The magnetic field strength of mpMRI magnetic resonance scanners commonly used in clinical practice is mostly 1.5T or 3.0T. The application of 3.0T magnetic resonance allows patients to no longer accept the use of rectal coils and makes the examination images clearer, making it the most commonly used magnetic field strength for mpMRI. The main problems of 3.0T prostate magnetic resonance examinations are low specificity (false positive results) and insufficient accuracy in determining tumor staging. At present, there is no research and exploration on the use of 5.0T magnetic resonance in the diagnosis of prostate cancer in the world. This study intends to analyze and compare the differences between 5.0TbpMRI and 3.0TbpMRI in the diagnosis of prostate cancer through a prospective, paired-design diagnostic trial, and try to explore whether 5.0TbpMRI can improve the limitations of 3.0TbpMRI in the diagnosis of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has at least one indication for prostate biopsy (Chinese expert consensus on prostate biopsy (2022 edition) );
2. The primary prostate cancer has no other cancer history;
3. The 3.0TbpMRI examination was completed, and the images were clear and accessible;
4. The 5.0TbpMRI examination was further completed, and the images were clear and accessible;
5. The patient fully understands the relevant content of the study and voluntarily signs the informed consent.

Exclusion Criteria:

1. The patient has contraindications to MRI examination, such as metal plates and heart stents in the body;
2. The patient does not have an indication for prostate biopsy or refuses biopsy;
3. The patient has contraindications to prostate biopsy;
4. 3.0T MRI considers that the patient has multiple lymph node or bone metastases;
5. The patient has undergone other prostatic surgery in the past;
6. The patient is unable to cooperate, has communication barriers, or refuses to sign the informed consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study mainly screened patients who need to complete mainly included serum PSA test, digital rectal examination, and 3.0TbpMRI and with indications of prostate biopsy. An informed consent conversation was conducted with the patient. After the patient fully understood the content of the study and signed the informed consent form, the researcher guided and arranged the 5.0TbpMRI examination throughout the process. All patients should complete the prostate biopsy according to the routine diagnosis and treatment process. The pathological diagnosis results of the prostate biopsy are the diagnostic gold standard of this study. The accuracy of 3.0TbpMRI and 5.0TbpMRI in preoperative prostate cancer tumor staging based on the final pathological results of radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the diagnostic efficacy of 5.0TbpMRI and 3.0TbpMRI for prostate cancer. | through study completion, an average of 1 month
  Definitions: csPCa, Gleason score ≥ 3+4， ISUP grade ≥ 2; agPCa, Gleason score ≥ 3+3， ISUP grade ≥ 1.
  Evaluation indexes: ROC curves and AUC value (95%CI) , Sensetivity, Specificity, Positive predictive value and negative predictive value.

SECONDARY OUTCOMES:
Evaluation of the reliability (repeatability) of the diagnostic test. | through study completion, an average of 1 month
  The inter-reader agreement was evaluated using Cohen's kappa analysis (Cohen's kappa coefficeint, P-value and 95%CI)
Comparative analysis of the accuracy of 5.0TbpMRI and 3.0TbpMRI in determining the stage of prostate cancer | through study completion, an average of 2 months
  Accuracy of prostate capsule invasion, seminal vesicle invasion and pelvic lymph node metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xiao, M.D., Principal Investigator — The First Affiliated Hospital of USTC
Locations (1):
- Department of Urology, The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided